CLINICAL TRIAL: NCT03355781
Title: Childhood Trauma in Schizophrenia: Exploration of Links Between Gene Expression, Cerebral Morphology and Symptomatology. SCHIZO' TRAUMA
Brief Title: Childhood Trauma in Schizophrenia: Exploration of Links Between Gene Expression, Cerebral Morphology and Symptomatology
Acronym: SCHIZO'TRAUMA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1608039; 2017-A00408-45 (Other: ANSM)
Record Dates: First submitted 2017-11-10; First posted 2017-11-28 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Schizophrenia
Keywords: childhood trauma; candidate gene expression; cerebral morphology; schizophrenic symptomatology; conceptual framework of stress vulnerability
MeSH Terms: conditions — Schizophrenia | interventions — Magnetic Resonance Imaging; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Schizophrenic patients: Patients will have clinical psychiatric evaluation, brain imaging and blood sample
  Interventions: Device: magnetic resonance imaging (MRI); Procedure: Blood sample; Other: Clinical psychiatric evaluation
- Related volunteers (first degree relative of patient): Related volunteers will have clinical psychiatric evaluation, brain imaging and blood sample
  Interventions: Device: magnetic resonance imaging (MRI); Procedure: Blood sample; Other: Clinical psychiatric evaluation
- Healthy volunteers: Healthy volunteers will have clinical psychiatric evaluation, brain imaging and blood sample
  Interventions: Device: magnetic resonance imaging (MRI); Procedure: Blood sample; Other: Clinical psychiatric evaluation

INTERVENTIONS:
Device: magnetic resonance imaging (MRI) — brain imaging : structural anatomy, emotional congruence, anatomic connectivity, functional connectivity
Procedure: Blood sample — 27,5 ml of blood sample : genetic analysis and biobank
Other: Clinical psychiatric evaluation — Global Assessment Scale(GAS),Mini International Neuropsychiatric Interview(MINI),Positive and Negative Symptoms Scale(PANSS),Family Interview for Genetic Studies(FIGS),Calgary Depression Scale for Schizophrenia(CDSS),extrapyramidal side effects evaluation or Simpson-Angus scale evaluation(ESRS),Apathy Evaluation Scale(AES-C),State-Trait Anxiety Inventory(STAI),Beck Depression Inventory(BDI-13),Eysenck Personality Questionnaire-Revised(EPQ-R),Assessment of Schizotypal Personality(SPQ),Emotion Regulation Questionnaire(ERQ),Emotional Reactivity Scale(ERS),Toronto Alexithymia Scale(TAS-20),social anhedonia scale(SAS),Childhood Trauma Questionnaire(CTQ),Clinical-administered Post Traumatic Stress Disorder Scale(CAPS),Wechsler Adult Intelligence Scale(WAIS-III),Trail Making Test(TMT),Pen and paper visuospatial working memory(DOT-test),impulsivity test(GoStop),Stroop test,National Adult Reading Test(NART),Wechsler Adult Intelligence Scale(WAIS-III),Facial Emotion Recognition task(FER)

SUMMARY:
Childhood trauma is known as a vulnerability factor in schizophrenia. In healthy volunteers, these adversities are linked to a decrease of grey matter of the brain, similar to those observed in schizophrenia.

In a previous study based on Voxel-Based Morphometry (VBM), including 21 schizophrenic patients and 30 healthy volunteers, the investigators shown a negative correlation between emotional neglect (important dimension in childhood trauma) and grey matter decrease. This strong correlation was significantly higher in schizophrenic patients than in healthy volunteers, suggesting a higher genetic predisposition to environmental factors in schizophrenic people.

Currently, interaction between genetic predisposition and environmental stress factors is the major model for understanding in schizophrenia. In order to analyze both effects on human body, particularly on brain, several studies currently focus on the product of genetic expression, the ribonucleic acid (ARN).

The purpose of this study is to provide an explanatory model of links between childhood trauma, candidate gene for schizophrenia expression, cerebral morphology and schizophrenic symptomatology. Using conceptual framework of stress vulnerability, structural equation modeling (SEM) will allow testing causal link between these different variables.

ELIGIBILITY:
Inclusion Criteria of patients :

* For women with reproductively active age period: suitable contraceptive method and negative pregnancy test
* Schizophrenia diagnosis (according to DSM 5)
* Regular follow-up care at hospital
* No change in antipsychotic medication (medication AND dosage) within at least six weeks
* Patient into remission : constant dosage, out-patient and meeting Andreassen criteria
* Who have given their informed consent before participating in the study.
* Physical examination without significant clinical physical anomaly
* No serious somatic pathology
* Affiliates or entitled to a social security scheme

Exclusion Criteria of patients :

* For women with reproductively active age period: no suitable contraceptive method (oral, hormonal, intramuscular, intrauterine device, or surgical)
* Pregnancy or breastfeeding
* Not meeting schizophrenic criteria according to DSM 5 or presenting resistant schizophrenic criteria according Kane criteria
* Presenting a serious somatic disorder or neurological (particularly Parkinson disease, epilepsy, tardive dyskinesia)
* Cardiovascular, hepatic or serious renal diseases
* Contraindication to MRI examination, particularly ocular or intracranial metallic foreign object,pacemaker, artificial heart valve, surgical clip
* Claustrophobia, significant tatoo in the high part of the body, IUD incompatible with MRI 3Tesla
* Alcohol or drug addiction, within the last year
* Recruited in other clinical trial or exclusion period from previous trial.
* Susceptibility to self-harm behaviour according to investigator

Inclusion Criteria of Related volunteers :

* Age, gender and socio-educational level similar to recruited patients
* Who have given their informed consent before participating in the study.
* First degree relative of schizophrenic patient diagnosed according DSM IV criteria
* No schizophrenia diagnosis according DSM IV criteria
* No psychiatric history and free of psychotropic drugs/treatment
* Physical examination without significant clinical anomaly
* Affiliates or entitled to a social security scheme

Exclusion Criteria of Related volunteers :

* For women with reproductively active age period: no suitable contraceptive method (oral, hormonal, intramuscular, intrauterine device, or surgical)
* Pregnancy or breastfeeding
* Presenting somatic, neurological or psychiatric disorder
* Alcohol or drug addiction, within the last year
* Recruited in other clinical trial or exclusion period from previous trial.
* Contraindication to MRI examination, particularly ocular or intracranial metallic foreign object, pacemaker, artificial heart valve, surgical clip
* Claustrophobia, significant tatoo in the high part of the body, IUD incompatible with MRI 3Tesla

Inclusion Criteria of Healthy volunteers :

* Age, gender and socio-educational level similar to recruited patients
* Who have given their informed consent before participating in the study.
* No schizophrenia diagnosis according DSM IV criteria
* No personal or family history of psychiatric disorders
* Free of psychotropic drugs/treatment
* Physical examination without significant clinical anomaly
* Affiliates or entitled to a social security scheme

Exclusion Criteria of Healthy volunteers :

Beside the absence of schizophrenia diagnosis, healthy volunteers should meet the same exclusion criteria as patients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Schizophrenic patients, related volunteers (first degree relative of patient) and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Childhood Trauma Questionnaire (CTQ) for childhood trauma. | 5 days
  development of an etiopathogenic model characteristic of schizophrenia
  Childhood Trauma Questionnaire : to assess five types of childhood trauma :
  1. Emotional neglect
  2. physical abuse
  3. emotional abuse
  4. physical neglect
  5. sexual abuse
  Each item being rated in 5 answer choice from 1 to 5 (never, rarely, sometimes, often or very often)
Quantitative measurement of RNAs | 5 days
  development of an etiopathogenic model characteristic of schizophrenia
Voxel-based morphometry (VBM) for total gray matter | 5 days
  development of an etiopathogenic model characteristic of schizophrenia
Voxel-based morphometry (VBM) for regional gray matter density. | 5 days
  development of an etiopathogenic model characteristic of schizophrenia

SECONDARY OUTCOMES:
Connectivity in the cortico-limbic circuit | 5 days
Volumetry of the brain | 5 days
Correlation of BOLD activity in the cortico-limbic circuit in patients with patients with symptomatic variables | 5 days
  symptomatic variables : PANSS scale
Correlation of BOLD activity in the cortico-limbic circuit with emotional variables | 5 days
  emotional variables : ERS scale, ERQ scale, TAS-20 scale, SAS scale, AES-C scale
Correlation of BOLD activity in the cortico-limbic circuit with personality characteristics | 5 days
  personality characteristics : EPQ-R scale, SPQ scale
Correlation of BOLD activity in the cortico-limbic circuit with history of trauma in childhood | 5 days
  history of trauma in childhood : CTQ scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No